CLINICAL TRIAL: NCT04759469
Title: Effect of Time-efficient Exercise Training on Cardiometabolic Risk Factors in Type II Diabetic Patients: A Randomized Mixed-methods Feasibility Study
Brief Title: Effect of Exercise on Cardiometabolic Risk Factors in Type II Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Hady Atef Labib, Lecturer of physical therapy for cardiopulmonary disorders, Faculty of Physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIIT on DM
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type II diabetes; cardiometabolic risk; high-intensity interval training
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval training (HIIT) (Experimental): A high-intensity interval training program for 3 days/week (day after day) for 12 weeks on atreadmill (Biodex RTM500, Biodex Inc., New York), with a gradual increase in the program intensity.
  Interventions: Behavioral: High-intensity interval training
- Moderate intensity interval training (MIIT) (Active Comparator): A moderate intensity interval training program for 3 days/week (alternate days) on a treadmill (Biodex RTM500, Biodex Inc., New York), with a gradual increase in the program.
  Interventions: Behavioral: Moderate intensity interval training

INTERVENTIONS:
Behavioral: High-intensity interval training — High-intensity interval training is a form of intermittent training using relatively high exercise intensity
  Arms: High-intensity interval training (HIIT)
Behavioral: Moderate intensity interval training — Moderate intensity interval training is a form of intermittent training using moderate exercise intensity
  Arms: Moderate intensity interval training (MIIT)

SUMMARY:
Background: Physical activity is known to modify some of the diabetes risk factors; however, solid evidence is still needed to precisely know the optimum form of training best fits the individual needs of type II diabetic (T2D) patients.

DETAILED DESCRIPTION:
Objectives: the purpose of this study was to compare between high intensity interval training (HIIT) and moderate-intensity interval training (MIIT) effect on functional capacity (as a cardiorespiratory parameter), and on glucose control and glycated hemoglobin (HbA1C) (as metabolic parameters) in T2D patients, and to test exercise acceptability within these patients. Methods: 60 participants had participated in this study. Their ages ranged from 45 to 65 years. They were randomized into two equal groups (30/group); group (A) did HIIT and group (B) did MIIT. Both groups received 12 weeks of training. Measurements for six minute walking distance (6MWD), fasting blood glucose (FBG), and HbA1C levels were done before and after the study. Physical activity enjoyment scale (PACES) were filled by the patients by the end of the study; testing exercise enjoyment.

ELIGIBILITY:
Inclusion Criteria:

* Controlled type 2 diabetic patients who were clinically stable for at least 3 months before entering the study,
* Aged 45-65 years
* Non-smokers
* body mass index (BMI) ranged between 20 to 39.9 Kg/m2
* Fasting blood glucose ranged from (126-160) mg/dl
* Sedentary lifestyle who didn't engage in physical activity for more than half an hour/ day for at least one month before entering the study.

Exclusion Criteria:

* unstable medical condition
* smoker, recent surgery
* Body mass index is more than 39.9 kg/m2 or less than 20 kg/m2
* Any known musculoskeletal or neurological conditions that might interfere with the execution or the assessment of the exercise

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
six minute walking distance (in meters) | 12 weeks
  represent aerobic capacity (distance walked in 6 min)
Glycated Hemoglobin (HbA1C) | 12 weeks
  Representing glucose control over 120 days
Fasting blood glucose | 12 weeks
  Representing glucose level after 9 hours fasting
Exercise enjoyment and acceptability | 12 weeks
  The Physical Activity Enjoyment Scale (PACES) score, out of 119. It is an 18-item scale that assesses enjoyment for physical activity by asking participants to rate "how you feel at the moment about the physical activity you have been doing" using a 7-point bipolar Likert scale, from 1 (I enjoy it) to 7 (I hate it). Eleven items were negatively worded and seven items were positively worded. After reverse scoring the 11negatively worded items, an overall enjoyment for physical activity score is determined by summing the items, with a range of 18-126 being possible. Higher scores indicate higher enjoyment.

SECONDARY OUTCOMES:
Adherence rates | 12 weeks
  To what extent the patients will adhere to the exercise protocol

CONTACTS AND LOCATIONS:
Overall Officials: Hady Atef, PhD, Study Director — Lecturer of physical therapy, Cairo University, Egypt
Locations (1):
- Alkasr Alaini hospital, Cairo, AI Qahirah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
After approval can be shared
Supporting Information: Study Protocol
Time Frame: after 1 month for12 months
Access Criteria: will upload it to the journal of publication